CLINICAL TRIAL: NCT00588315
Title: In Vivo Confocal Microscopy of Cutaneous Neoplasms and Normal Skin
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 99-099
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- skin lesions: The integrated dermoscopic-and-confocal microscopic video-mosaics will be used to compare morphologic patterns and cellular patterns to each other and to the corresponding pathology
- normal skin: The integrated dermoscopic-and-confocal microscopic video-mosaics will be used to compare morphologic patterns and cellular patterns to each other and to the corresponding pathology

SUMMARY:
The purpose of this study is to investigate new non-invasive imaging techniques for the evaluation of skin lesions, as well as normal skin. Our primary goal is to collect and study these images of different skin lesions along with matching biopsy specimens. The long-term goal is to develop a technique that will improve the early detection of skin cancer and eliminate the need for many skin biopsies.

The High-resolution OCT (Apollo Medical Optics) device can provide both cross-sectional and en-face images with cellular information. Real-time color images through the same objective with OCT are also provided to show the OCT imaging location of lesion. The color image can be registered simultaneously on a larger dermoscopic image obtained by an external dermoscope. The imaging mode of cross-sectional, en-face and color image can be switched arbitrarily to align the lesion and obtain high-resolution images efficiently. The total imaging time is around 10 to 15 minutes depending on the number of images to be obtained.

To help identify more diagnostic features of optical imaging and better understand their histology correlation, we have developed a novel technique called "precision biopsy". Precision biopsy is an optical imaging guided, feature-targeted mini-biopsy. Once the feature of interest is identified and isolated by the optical imaging, a 2.0 mm punch biopsy is performed. Besides cosmetic benefit of minimal scarring, this tissue sparing biopsy captures the "feature of interest" for histology revelation.

Additionally, the histologic features of precision biopsy will be compared to images gathered by multi-modal optical imaging. The precision biopsy will also be compared to the traditional shave biopsy or shave excision, to determine whether the diagnostic information is comparable between the two methods.

For live remote control (LRC) imaging consultation, MSK dermatologist will based on his clinical examination. An imaging technician will perform the clinical and dermoscopic imaging, while the expert reader will perform confocal imaging remotely via a HIPPA compliant Webex platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than or equal to 10 years of age.
* Patients with a skin lesion with anticipated epidermal and superficial dermal histologic alterations amenable to visualization by surface confocal microscopy.
* Healthy volunteer subjects older than or equal to 10 years old.
* Ability to give informed consent.

Exclusion Criteria:

* Patients who are allergic to fluorescein sodium.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the Dermatology, Clinical Immunology Services, Pediatrics and Radiology Oncology departments that are determined to have a skin lesion with anticipated epidermal and superficial dermal histologic alterations amenable to visualization by surface confocal microscopy will be offered the opportunity to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1889 (Actual)
Dates: Start 1999-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The study is a descriptive one. No formal statistical testing of correlations will be performed. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manu Jain, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Hauppauge (Consent only), Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm